CLINICAL TRIAL: NCT00010699
Title: Effect of High Dose Vitamin E on Carotid Atherosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000005-02 (NIH); NCT00009373 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Diseases
Keywords: cvd
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Vitamin E

INTERVENTIONS:
Drug: Vitamin E

SUMMARY:
The primary aim of the present study is to test the effect of alpha-tocopherol supplementation on the progression of carotid atherosclerosis in patients with coronary artery disease

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of morbidity and mortality in Westernized populations. Oxidation of low-density lipoprotein (LDL) appears to be a crucial step in atherogenesis. Thus, the role of dietary micronutrients in decreasing LDL oxidation assumes considerable significance. The most consistent data with respect to micronutrient antioxidants and atherosclerosis appear to relate to a-tocopherol (AT), the predominant lipid-soluble antioxidant in LDL. In addition to decreasing LDL oxidation, data support an effect of AT on critical cells in atherogenesis (monocytes, smooth muscle cells, and endothelium) that are potentially anti-atherogenic.

The primary aim of the present study is to test the effect of AT supplementation (1200 IU/day of RRR-AT) in a placebo-controlled, randomized double blind trial over 2 years on the progression of carotid atherosclerosis in patients with coronary artery disease (stable angina pectoris or previous myocardial infarction).

Subjects recruited would have to be on the American Heart Association Phase II diet and a HMG CoA reductase inhibitor for at least one year and have an LDL cholesterol <125 mg/dL on 2 visits at least 4 weeks apart during the 10 month lead in phase. Intimal-medial thickness (IMT) of both carotids, including the common carotid, the bulb and the proximal internal carotid will be determined by high-resolution B-mode sonography. At six month intervals blood samples will be obtained for liver enzymes, creatinine, complete blood count, lipid profile, antioxidant and fatty acid levels, LDL oxidation, plasma soluble CAMS (cell adhesion molecules) and monocyte activity. Also, an early morning urine sample will be obtained for F2 -isoprostanes, a direct measure of lipid peroxidation. IMT will be determined at baseline, 1, 1.5 and 2 years. The mean change in IMT and rate of progression will be compared between the AT and placebo groups. Following isolation, the LDL will be subjected to copper catalyzed oxidation over a 5-hour period. From this will be obtained the lag phase and oxidation rate. Isolated monocytes will be activated with lipopolysaccharide and the following activities assayed: superoxide anion release, interleukin-1 j3 release and adhesion to human endothelium. F2 isoprostanes and VCAM, ICAM, and E- 8 P-Selectin will be quantitated by ELISA. AT levels and the parameters of LDL oxidation and monocyte activity will be correlated with changes in IMT.

If this study shows that high-dose AT supplementation is beneficial in retarding atherosclerosis this could emerge as an important adjunctive therapy in the management of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Must be on the American Heart Association Phase II diet and a HMG CoA reductase inhibitor for at least one year
* Have an LDL cholesterol <125 mg/dL on 2 visits at least 4 weeks apart during the 10 month lead in phase.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ishwarlal Jialal, MD, Ph.D., Principal Investigator — Department of Pathology
Locations (2):
- United States (2):
  - UC Davis Medical Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California